CLINICAL TRIAL: NCT06003400
Title: Proof of Concept Open Label, Clinical Trial to Evaluate the Safety and Efficacy of the "FITT" Device in Diabetic Foot Ulcers Patients
Acronym: TriO FITT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri.O Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-21-01
Record Dates: First submitted 2023-07-25; First posted 2023-08-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Physical Examination; Vital Signs

STUDY DESIGN:
Intervention Model Description: Administration of Tri.O FITT for upto 12 weeks or until wound closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tri.O FITT (Experimental): The study patients will undergo a screening period of upto 4 weeks, a traetment period of upto 12 weeks and a follow-up period of upto 12 additional weeks.
  Interventions: Device: Study treatment administration (TriO FITT); Diagnostic Test: Physical Examination; Diagnostic Test: Vital Signs; Diagnostic Test: Hematology Blood Tests; Diagnostic Test: Biochemistry Blood Test; Diagnostic Test: Wound Digital Photography; Diagnostic Test: Urine pregnancy test; Other: Visual Analogue Scale; Other: SF-36; Diagnostic Test: Wounds evaluation

INTERVENTIONS:
Device: Study treatment administration (TriO FITT) — Patients will be treated with the study device 2-3 times per week (determined by their wagner score) for an hour at each visit. treatment will include a combination of methods (the exact details is patented by the company and can not be elaborated).
Diagnostic Test: Physical Examination — physical examination will include an overall examination of the patient's body for any iregular findings and or physical changes from baseline.
Diagnostic Test: Vital Signs — vital signs measurement will include blood pressure, pulse and oral temperature as well as hight and weight.
Diagnostic Test: Hematology Blood Tests — complete CBC, coagulogram (PT, aPTT); D-dimer; C-reactive protein;; Ferritin; fibrinogen,
Diagnostic Test: Biochemistry Blood Test — urea, creatinine, uric acid, sodium, potassium, chloride, calcium, glucose, glycated hemoglobin, alkaline phosphatase (FA), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin and fractions ( BTF), total proteins and fractions (PTF), lipid profile (total cholesterol, fractions and triglycerides).
Diagnostic Test: Wound Digital Photography — 3 photographs of the wound taken before wash, after wash and after treatment.
Diagnostic Test: Urine pregnancy test — for women with childbearing potential
Other: Visual Analogue Scale — Visual Analogue Scale - visual scale scoring 1-10 measuring pain, 10 being worst pain.
Other: SF-36 — SF-36 - quality of life questionnaire scaling from 0-100, 100 being best quality of life.
Diagnostic Test: Wounds evaluation — including size measurements and visual description.

SUMMARY:
The TriO FITT device is designed to improve the symptoms of chronic diabetic ulcers.

The mechanism of action of the device optimizes and combines the administration known supproting treatments to chronic diabetic ulcers. The treatment is astimated to improve the wound conditions of acute and chronic diabetic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-80 years old
* Chronic Diabetes Mellitus type 1 and type 2 diagnosed at least 3 years before the screening
* Have a single non-infected diabetic hard-to-heal wound (ulcers/foot ulcers) ≤ 0.8-40 cm2 wound area at start of treatment, for period of at least for 3 months.
* Wagner classification stage 1 or 2 or post-debridement stage 3.
* At least moderate blood perfusion into the affected limb as defined by Ankle Brachial Index (ABI) ≥0.65
* Stable diabetic drugs 4 weeks before Screening
* Be available for the entire study period, and be able and willing to adhere to protocol requirements
* Provide written informed consent prior to admission into the study

Exclusion Criteria:

* Have a glycosylated hemoglobin (HbA1c) > 10.5%
* Have more than one wound
* Have a body mass index (BMI) > 40 kg/m2
* Have visible bone exposure at wound site
* Anemia (Hemoglobin < 9 g/dL) or White Blood Cells count > 11,000/μL or Platelets count < 100,000/μL or liver function tests > 3 times upper normal lab values or Creatinine > 3 mg/dL; any indication of malnourishment (Albumin < 3 g/dL); INR>2 or any other clinically significant blood and urinalysis tests per the physician's discretion
* Patients with unstable hypertension
* Have any clinically significant chronic or acute illness during the 4 weeks prior to admission into the study, except diabetes type 1 or 2 or during screening period
* Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years, not using a medically approved method of contraception (i.e., oral, transdermal, or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterility), or females who test positive on a urine-based pregnancy test
* Participation in a clinical study or use of an investigational drug within 30 days prior to admission to this study
* Patients with active Gangrenous foot ulcers
* Active osteomyelitis (Have any signs of infection in the wound (which could be linked to raised body temperature), abscess, cellulitis, necrosis, erythema, mild drainage or known osteomyelitis)
* Patients with uncontrolled hyperthyroidism
* Patients with history of collagen diseases
* Patients with known allergy to ozone
* Anxiety, Depression, history of Mental illness or patient under Guardian
* Any medical condition for which the investigator deems the subject unable to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Safety measured by number of patients who lack adverse events throughout the study. | 0 to 28 weeks
Change in pain level between visits 1 and the last treatment evaluated by VAS scale | 0 to 28 weeks
  pain levels will be measured by the precent of change in VAS pain raiting scale.
Change in Quality of life (QoL) between visits 1 and the last treatment, measured by SF-36 | 0 to 28 weeks
  score measures from 0 to 100, 100 being good quality of life.
Change in wound size between V1 and the last treatment | 0 to 28 weeks
  change in size (cm^2)

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Ben Ari, Study Director — CEO
Locations (1):
- Hilel Yafe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No